CLINICAL TRIAL: NCT00171028
Title: A Double-Blind, Randomized, Multi-Center Study Followed By 12 Months Open-Label Treatment To Evaluate The Dose Response And Safety Of Valsartan In Pediatric Hypertension Patients 1 - 5 Years Of Age
Brief Title: A Study Of Valsartan Used To Treat Hypertension For Up To 56 Weeks In Children Ages 1 - 5 Years Who Have Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CVAL489A2307
Record Dates: First submitted 2005-09-10; First posted 2005-09-15 (Estimated); Last update posted 2011-11-08 (Estimated); Status verified 2006-06

CONDITIONS: Hypertension
Keywords: PEDIATRIC HYPERTENSION; PEDIATRIC; VALSARTAN
MeSH Terms: conditions — Hypertension | interventions — Valsartan

INTERVENTIONS:
Drug: valsartan

SUMMARY:
Drugs used to treat hypertension in adults should also be effective in treating high blood pressure in infants and children. This study will test the safety and efficacy of valsartan in lowering blood pressure in children 1 - 5 years old whose parents grant permission to participate.

ELIGIBILITY:
Inclusion Criteria:

* CHILDREN HAVE BLOOD PRESSURE LEVEL =>95TH PERCENTILE FOR AGE,GENDER & HEIGHT
* PARENTAL CONSENT MUST BE GRANTED

Exclusion Criteria:

* BLOOD PESSURE IS =>25% HIGHER THAN 95TH PERCENTILE FOR AGE, GENDER & HEIGHT
* SERIOUS, CLINICALLY SIGNIFICANT FINDINGS UPON EXAMINATION AND LABORATORY OR OTHER ASSESSMENTS

Other protocol-defined exclusion criteria will apply.

Ages: 1 Year to 5 Years | Sex: All
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2003-12; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline systolic blood pressure after 2 and 4 weeks

SECONDARY OUTCOMES:
Change from baseline systolic blood pressure after 4 weeks
Change from baseline diastolic blood pressure after 2 weeks
Change in 2 week diastolic blood pressure after 2 more weeks
Change in baseline diastolic blood pressure after 4 weeks
Adverse events, serious adverse events, and laboratory values during 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Pharmaceuticals, East Hanover, New Jersey, United States

REFERENCES:
- [Derived] Flynn JT, Meyers KE, Neto JP, de Paula Meneses R, Zurowska A, Bagga A, Mattheyse L, Shi V, Gupte J, Solar-Yohay S, Han G; Pediatric Valsartan Study Group. Efficacy and safety of the Angiotensin receptor blocker valsartan in children with hypertension aged 1 to 5 years. Hypertension. 2008 Aug;52(2):222-8. doi: 10.1161/HYPERTENSIONAHA.108.111054. Epub 2008 Jun 30. PMID 18591457